CLINICAL TRIAL: NCT02404701
Title: Effect of Over-the-counter Dietary Supplements on Kidney Stone Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-0076
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Hyperoxaluria
MeSH Terms: conditions — Hyperoxaluria | interventions — Tea; Vaccinium myrtillus extract; milk-thistle extract; Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Aloe vera with cactus (Experimental): 1 capsule (500 mg), 2 times/day
  Interventions: Dietary Supplement: Aloe vera with cactus
- Cranberry (Experimental): 3 capsules (810 mg), 2 times/day
  Interventions: Dietary Supplement: Cranberry
- Green tea extract (Experimental): 2 capsules (630 mg), 2 times/day
  Interventions: Dietary Supplement: Green tea extract
- Bilberry (Experimental): 1 softgel (1000 mg), 2 times/day
  Interventions: Dietary Supplement: Bilberry
- Cinnamon (Experimental): 1 capsule (500 mg), 2 times/day
  Interventions: Dietary Supplement: Cinnamon
- Milk thistle (Experimental): 1 capsule (250 mg), 3 times/day
  Interventions: Dietary Supplement: Milk thistle
- Turmeric (Experimental): 1 capsule (450 mg turmeric + 50 mg turmeric extract), 1 time/day
  Interventions: Dietary Supplement: Turmeric
- Aloe vera (Experimental): 1 capsule (470 mg), 2 times/day
  Interventions: Dietary Supplement: Aloe vera

INTERVENTIONS:
Dietary Supplement: Aloe vera with cactus — Eligible participants who provide consent/authorization will report for an orientation visit (1 of 3 visits), during which participants will: provide a medical history and a 24-hour diet recall, have height and weight measured, learn how to collect 24-hour urine, receive instructions on following a standardized diet for 7 days, learn to use a food scale and provide diet records, and receive a 4-day supply of the supplement they were allocated to take along with instructions. After 3 days on the diet (no supplement), participants will return their first (of 2) diet record and 24-hour urine collection. After 4 days on the diet while taking the supplement, participants will return their second (and final) completed diet record and their second (and final) 24-hour urine collection.
  Other Names: Walgreens
  Arms: Aloe vera with cactus
Dietary Supplement: Cranberry — Eligible participants who provide consent/authorization will report for an orientation visit (1 of 3 visits), during which participants will: provide a medical history and a 24-hour diet recall, have height and weight measured, learn how to collect 24-hour urine, receive instructions on following a standardized diet for 7 days, learn to use a food scale and provide diet records, and receive a 4-day supply of the supplement they were allocated to take along with instructions. After 3 days on the diet (no supplement), participants will return their first (of 2) diet record and 24-hour urine collection. After 4 days on the diet while taking the supplement, participants will return their second (and final) completed diet record and their second (and final) 24-hour urine collection.
  Other Names: Puritan's Pride
  Arms: Cranberry
Dietary Supplement: Green tea extract — Eligible participants who provide consent/authorization will report for an orientation visit (1 of 3 visits), during which participants will: provide a medical history and a 24-hour diet recall, have height and weight measured, learn how to collect 24-hour urine, receive instructions on following a standardized diet for 7 days, learn to use a food scale and provide diet records, and receive a 4-day supply of the supplement they were allocated to take along with instructions. After 3 days on the diet (no supplement), participants will return their first (of 2) diet record and 24-hour urine collection. After 4 days on the diet while taking the supplement, participants will return their second (and final) completed diet record and their second (and final) 24-hour urine collection.
  Other Names: Puritan's Pride
  Arms: Green tea extract
Dietary Supplement: Bilberry — Eligible participants who provide consent/authorization will report for an orientation visit (1 of 3 visits), during which participants will: provide a medical history and a 24-hour diet recall, have height and weight measured, learn how to collect 24-hour urine, receive instructions on following a standardized diet for 7 days, learn to use a food scale and provide diet records, and receive a 4-day supply of the supplement they were allocated to take along with instructions. After 3 days on the diet (no supplement), participants will return their first (of 2) diet record and 24-hour urine collection. After 4 days on the diet while taking the supplement, participants will return their second (and final) completed diet record and their second (and final) 24-hour urine collection.
  Other Names: Puritan's Pride
  Arms: Bilberry
Dietary Supplement: Cinnamon — Eligible participants who provide consent/authorization will report for an orientation visit (1 of 3 visits), during which participants will: provide a medical history and a 24-hour diet recall, have height and weight measured, learn how to collect 24-hour urine, receive instructions on following a standardized diet for 7 days, learn to use a food scale and provide diet records, and receive a 4-day supply of the supplement they were allocated to take along with instructions. After 3 days on the diet (no supplement), participants will return their first (of 2) diet record and 24-hour urine collection. After 4 days on the diet while taking the supplement, participants will return their second (and final) completed diet record and their second (and final) 24-hour urine collection.
  Other Names: Puritan's Pride
  Arms: Cinnamon
Dietary Supplement: Milk thistle — Eligible participants who provide consent/authorization will report for an orientation visit (1 of 3 visits), during which participants will: provide a medical history and a 24-hour diet recall, have height and weight measured, learn how to collect 24-hour urine, receive instructions on following a standardized diet for 7 days, learn to use a food scale and provide diet records, and receive a 4-day supply of the supplement they were allocated to take along with instructions. After 3 days on the diet (no supplement), participants will return their first (of 2) diet record and 24-hour urine collection. After 4 days on the diet while taking the supplement, participants will return their second (and final) completed diet record and their second (and final) 24-hour urine collection.
  Other Names: Puritan's Pride
  Arms: Milk thistle
Dietary Supplement: Turmeric — Eligible participants who provide consent/authorization will report for an orientation visit (1 of 3 visits), during which participants will: provide a medical history and a 24-hour diet recall, have height and weight measured, learn how to collect 24-hour urine, receive instructions on following a standardized diet for 7 days, learn to use a food scale and provide diet records, and receive a 4-day supply of the supplement they were allocated to take along with instructions. After 3 days on the diet (no supplement), participants will return their first (of 2) diet record and 24-hour urine collection. After 4 days on the diet while taking the supplement, participants will return their second (and final) completed diet record and their second (and final) 24-hour urine collection.
  Other Names: Puritan's Pride
  Arms: Turmeric
Dietary Supplement: Aloe vera — Eligible participants who provide consent/authorization will report for an orientation visit (1 of 3 visits), during which participants will: provide a medical history and a 24-hour diet recall, have height and weight measured, learn how to collect 24-hour urine, receive instructions on following a standardized diet for 7 days, learn to use a food scale and provide diet records, and receive a 4-day supply of the supplement they were allocated to take along with instructions. After 3 days on the diet (no supplement), participants will return their first (of 2) diet record and 24-hour urine collection. After 4 days on the diet while taking the supplement, participants will return their second (and final) completed diet record and their second (and final) 24-hour urine collection.
  Other Names: Puritan's Pride
  Arms: Aloe vera

SUMMARY:
The purpose of this study is to ascertain whether certain supplements promote excessive urinary oxalate excretion and increase the risk for calcium oxalate kidney stones. Supplements that enhance urinary oxalate excretion, as a result of their oxalate concentration or from some other mechanism (e.g., providing substrate for oxalate biosynthesis) will be identified by the investigators.

DETAILED DESCRIPTION:
The investigators hypothesize that certain over-the-counter dietary supplements will increase urinary excretion of oxalate as measured in 24-h urine collections. The investigators further hypothesize that the concentration of oxalate in dietary supplements may not be associated with urinary oxalate excretion, suggesting that other nutritional components of the supplements may be exerting an influence over oxalate biosynthesis, oxalate absorption in the gastrointestinal tract, and/or renal oxalate handling. These other factors include the form of oxalate in the supplement (water- vs. non water-soluble) and the supplement's concentration of ascorbic acid.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, no prior personal history of kidney stones

Exclusion Criteria:

* Personal history of kidney stones (by subjects' report); known allergy to any of the dietary supplements to be used in the study (by subjects' report); short bowel; active ulcerative colitis or irritable bowel disease; Crohns or Celiac disease; renal tubular acidosis; current use of topiramate or other carbonic anhydrase inhibitor, steroids, allopurinol, thiazide diuretics, or supplemental ascorbic acid >250 mg/day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Within-subject change in 24-hour urinary oxalate excretion from before and after supplementation | 7 days
  24-hour urine samples will be analyzed for oxalate by ion chromatography. The difference in oxalate between the baseline (non-supplement) and supplement phase will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina L Penniston, PhD, RD, Principal Investigator — Department of Urology, University of Wisconsin School of Medicine and Public Health
Locations (1):
- Department of Urology, School of Medicine & Public Health, University of Wisconsin, Madison, Wisconsin, United States